CLINICAL TRIAL: NCT05092854
Title: The Effect of AMP Human Sodium Bicarbonate Lotion on Physiological and Cognitive Performance During Dehydrated Heat Stress
Brief Title: The Effect of AMP Human Sodium Bicarbonate Lotion on Dehydrated Heat Stress
Acronym: AMP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: AMP Human; Park City, UT (Unknown); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Douglas J Casa, Principal Investigator, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H21-0054
Record Dates: First submitted 2021-09-26; First posted 2021-10-26 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Fluid Retention; Sodium Retention; Heat Stress; Dehydration (Physiology); Renal Injury; Electrolyte and Fluid Balance Conditions
Keywords: Sodium Bicarbonate; Amino Acid Supplementation; Topical Lotion; Renal Injury
MeSH Terms: conditions — Hypernatremia; Heat Stress Disorders; Dehydration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PR Lotion Topical Solution (Active Comparator): Dose Dependent Response: Different doses relative to the participant's body weight will be provided for provision onto the skin before beginning data collection procedures. The 'larger' dose will be composed of 0.8g/kg of the PR Lotion while the 'smaller' dose will be composed of 0.4g/kg of the PR Lotion. Participants will be instructed to apply the lotion primarily to their lower extremities and upper extremities as needed. This lotion will be applied once during the Intervention session of each phase completed and will remain on the skin for approximately 3.5 hours.
  Interventions: Other: PR Lotion - AMP Human Performance
- Placebo Lotion Topical Solution (Placebo Comparator): A dose of lotion relative to the participant's body weight will be provided for provision onto the skin before beginning data collection procedures. This dose will be approximately 0.8g/kg of the Placebo Lotion. Similar to the PR Lotion, participants will be instructed to apply the lotion primarily to their lower extremities and upper extremities as needed. This lotion will be applied once during the Intervention session of each phase completed and will remain on the skin for approximately 3.5 hours.
  Interventions: Other: Placebo Lotion
- Hydration Status (Experimental): Participants will be asked to partake in 5 total Intervention trials. Upon arrival to each trial, the participant will be asked to complete an 18-24 fluid restriction protocol to ensure their arrival within a dehydrated state. Depending on the phase randomization assigned to each participant, they will either be provided fluids to consume that will bring them back to an estimated level of 1% dehydration (total of 3/5 trials completed) or they will not be given any fluids to consume during the duration of the trial (total 2/5 trials completed). Participants will be considered completed with project participation upon the completion of each of the five trials outlined.
  Interventions: Other: PR Lotion - AMP Human Performance; Other: Placebo Lotion; Other: AminoVital - Rapid Recovery; Other: Placebo Supplement
- aminoVITAL - Amino Acid Rehydration Supplement (Active Comparator): Participants will be provided with 3 servings of a commercially available amino acid rehydration supplement for consumption after the completion of the dehydrated heat stress intervention. Participants will be instructed to consume each serving in a time-dependent manner over the 24-hour period after dismissal from the laboratory after completion of the Intervention session.
  Interventions: Other: AminoVital - Rapid Recovery
- Placebo Drink Supplement Solution (Placebo Comparator): Participants will be provided with 3 servings of a placebo rehydration supplement for consumption after the completion of the dehydrated heat stress intervention. Participants will be instructed to consume each serving in a time-dependent manner over the 24-hour period after dismissal from the laboratory after completion of the Intervention session.
  Interventions: Other: Placebo Supplement

INTERVENTIONS:
Other: PR Lotion - AMP Human Performance — Sodium Bicarbonate Topical Solution. For use of the PR Lotion solution, consumers are instructed to apply the lotion to areas of the body that have been identified as most likely to use during their activity (i.e. calves and thighs for runners, shoulders and forearms for swimmers, etc.). Moreover, the product can be applied up to 2 hours prior to beginning a workout or event with one use supporting a 4-6 hour workout. AMP Human has also verified the safety of their product as being well tolerated in consumers >2 years of age unless there is a known allergy to an ingredient on the label. Moreover, to the company's knowledge no side effects have been reported per the SAFETY Section at https://amphuman.com/pages/faq.
  Other Names:
  NDC Code: 72358-101-01 NDC Code: 72358-101-02 NDC Code: 72358-101-03
  Other Names: NDC Code: 72358-101-01; NDC Code: 72358-101-02; NDC Code: 72358-101-03
  Arms: Hydration Status; PR Lotion Topical Solution
Other: Placebo Lotion — Placebo Topical Solution. Lotion will be created by the AMP Human Performance company and will include all ingredients similar to the PR Lotion product except for the exclusion of sodium bicarbonate.
  Arms: Hydration Status; Placebo Lotion Topical Solution
Other: AminoVital - Rapid Recovery — AminoVITAL Rapid Recovery is a commercially available supplement that is not currently regulated by the FDA but does complete both internal quality control and third-party testing for all of their products. AminoVITAL Rapid Recovery has been certified by the Banned Substance Control Group (BSCG; https://www.bscg.org/certified-drug- free-supplements/?AminoVITAL) and has been certified to be free of 496+ drugs including WADA Prohibited Substances as well as prescription, over the counter, and illicit drugs not banned in sport. AminoVITAL Rapid Recovery is safe to consume multiple times within a single day and has been found most effective when taken within 30 minutes of cessation of exercise. No known side effects are associated with the ingestion of aminoVITAL Rapid Recovery; however, side effects of amino acid toxicity include gastrointestinal distress, nausea and headache.
  Arms: Hydration Status; aminoVITAL - Amino Acid Rehydration Supplement
Other: Placebo Supplement — Supplement will be created by the aminoVITAL company and will include all ingredients similar to the commercially available Rapid Recovery product except for the exclusion of the amino acid blend.
  Arms: Hydration Status; Placebo Drink Supplement Solution

SUMMARY:
The primary purpose of the proposed study is to evaluate the effects of a topical sodium bicarbonate lotion (PR Lotion, AMP Human, Park City, UT) on measures of hydration status and fluid balance in humans when exposed to the heat while resting and during light/moderate aerobic exercise. A secondary purpose is to examine these same effects with two differing dosage patterns of the lotion. A tertiary purpose is to investigate the effect of an amino acid rehydration beverage in comparison to a placebo on measurements of hydration, subjective assessments of stress, and vestibular as well as musculoskeletal measures of fatigue for up to 24-hours after the completion of both passive and exertional heat stress within a dehydrated state.

DETAILED DESCRIPTION:
Design This laboratory study will involve the inclusion of 20 male participants from the local community and university who are within the age range of 18 - 45 years old and can be classified as recreationally active adults as indicated by a VO2max minimum (45 ml/kg/min) who choose to volunteer for this research study. This project will be conducted within the thermal physiology laboratory, complete with a climatic chamber (Cantrol, CES +13/+44) located within the Human Performance Laboratory (HPL) at the University of Connecticut. We expect data collection to take approximately 3-4 months for completion and each interested individual will complete all five trials included within the study design within a randomized, counterbalanced order.

Participants will be randomly assigned de-identified codes, trial grouping orders, and allocation of amino acid rehydration beverages (i.e., aminoVITAL Rapid Recovery or Placebo) after approval has been provided and consent has been obtained. The order of participation will be counterbalanced between participants to ensure that there is not an order effect with each participant completing all 5 trials outlined in the study design. Additionally, for the post trial amino acid rehydration portion of the study only, participants will be matched based on an assortment of physiological variables measured (i.e., physical fitness [VO2max], body mass index, body surface area, age, height, and/or weight) in regards to their assigned allocation of the amino acid rehydration beverages (i.e., aminoVITAL Rapid Recovery or Placebo) that will be consumed during the recovery period of the study design.

Environmental Conditions Session I as well as all Baseline Visits and matched-control 24-hour Rehydration Sessions (i.e., AminoVITAL Rapid Recovery or Placebo) will be completed within thermoneutral conditions. Moreover, all Dehydration Periods associated with completion of the study will be completed by the participant outside of the laboratory. Finally, all counterbalanced testing sessions (i.e., 0.8PR-Fluid, 0.4PR-Fluid, PLA-Fluid, 0.8PR-Dry, and PLA-Dry) will be conducted within the climatic chamber set to a climate with an ambient temperature at approximately 330C (91.40F) and relative humidity at approximately 25%.

Baseline and VO2max Testing - Session 1 Session 1 will serve as a baseline testing session to obtain an assortment of physiological, vestibular, strength, and cognitive measurements to conduct an effective baseline measurement for each individual participating in this study. Physiological assessments will include measurements of each individual's body composition (height, weight, and body fat percentage), cardiovascular health (resting blood pressure, heart rate, and HRV), and aerobic fitness level via assessment of maximal oxygen consumption (VO2max). Furthermore, participants will be assessed for their cognitive abilities (ANAM testing battery), vestibular performance (BESS) and physical performance (grip strength and grip endurance). For the completion of this testing session, participants will be instructed to consume an efficient amount of fluids to ensure proper hydration for testing. Additionally, participants will be instructed to refrain from eating or smoking for up to 3 hours before the beginning of their session.

Arrival Procedures:

Upon arrival, subjects will be asked if they have refrained from excluded nutritional supplementation for the last 48 hours, exercise and alcohol consumption in the past 24 hours, and caffeine for the last 12 hours. Next, subjects will provide their nude body mass and a urine sample within a clean urine cup for the assessment of urine specific gravity (USG) and urine color to determine hydration status. Privacy will be afforded for each participant while obtaining body mass measures by taking measurements with the participant alone in a private room and the research team member reading the scale outside of the room. Those with a USG <1.020 will be allowed to proceed with the exercise protocol. Those with a USG between 1.020-1.025 will be given approximately 500ml of water for immediate consumption with the completion of an additional USG assessment to ensure participants are efficiently hydrated. Those with a USG >1.025 will be rescheduled for another day due to inadequate hydration. Upon completion participants will have their height measured via stadiometer and body composition assessed via air displacement plethysmography (BodPod®; Cosmed, Software Version 4.2+, Concord, CA, USA).

Testing Procedures:

Upon completion of all arrival procedures, participants will then be asked to don a heart rate strap and rest for approximately five minutes before having baseline cardiovascular measurements completed including resting heart rate variability (HRV), resting heart rate (HR), and blood pressure (BP). Afterwards, participants will then be asked to complete the baseline measurement for their cognitive performance battery which will include the completion of the Modified Balance Error Scoring System (BESS), hand grip strength and endurance and the ANAM testing battery. Afterwards, participants will then be asked to complete a maximal oxygen uptake (VO2max) test performed via running on a motorized treadmill within a thermoneutral environment. This assessment will be completed as a baseline assessment for the participant's aerobic fitness (VO2max test) and the results (i.e., minimum VO2max of 45 ml/kg/min) will be used as a final inclusionary criteria measurement for the participant. Please see the Measurements Completed section for further information regarding procedures completed when conducting these testing protocols.

Testing of Biomedical Intervention - Climatic Chamber Testing Sessions Participants will be eligible to initiate the testing phase of their participation approximately 48 hours after the completion of all Session 1 baseline protocols. Furthermore, a minimum of 72 hours (approximately 3 days) must pass between the completion of each testing session completed. However, participants will be provided flexibility in scheduling through the option to reschedule testing sessions if needed to accommodate their personal schedules or rescheduling within the laboratory space. As previously outlined, the order of trials completed will be randomized to limit the possibility of an order effect for responses obtained to be detected. Each trial will include a predetermined amount (i.e., 0.8g/kg or 0.4g/kg) of the biomedical intervention (PR lotion or Placebo lotion) to be provided by the project sponsor. Differential amounts will be provided to investigate if a dose-dependent response may be elicited for the benefits of application regarding the biomedical intervention. For all trials, participants will undergo fluid restriction to attain hypohydration. Moreover, participants will arrive to the laboratory in a dehydrated state (protocols regarding this have been provided further below) and will either receive a pre-determined fluid bolus to replace a portion of their previous day's losses (relative to their body composition) or no fluid. This will allow us to assess the efficiency of the biomedical intervention for the retention of fluids consumed during their exposure to both passive and exertional heat stress while in a dehydrated state.

Baseline Visits and Dehydration Periods To properly induce dehydration within study participants, they will be asked not to take in fluid or high fluid containing foods (i.e., soup, cereal with milk, etc.) for approximately 18-24 hours prior to their scheduled Climatic Chamber Testing Session. However, before the initiation of this fluid restriction period, participants will be asked to arrive to the HPL for the completion of a pre-testing Baseline Visit that will need to be conducted before the beginning of each individual phase within the study. This session will include the collection of the participant's nude body weight in addition to a spot urine sample and a blood draw. The collection of the participant's nude body weight and urine sample will be conducted within the privacy of a restroom within the HPL. Additionally, a single blood draw will be conducted for the collection of approximately 11 mL (~0.75 tablespoon) of blood. These measurements will be collected in order to provide a euhydrated baseline measurement to compare to the measurements collected at the beginning of each Climatic Chamber Testing Session to confirm that proper dehydration has been attained. At the completion of all the previously described tasks associated with this visit, participants will be provided a urine jug for the collection of a 24-hour urine sample which will be provided to the administrating research personnel upon arrival for their upcoming testing session. Additionally, participants will also be asked to consume a similar dietary intake between each lab visit (measured via completion of the dietary recall log), with the exception of fluid and high fluid containing foods. This time period has been designed to elicit an

~1.5-3.0% loss in body mass and has been performed previously in our laboratory (See UCONN IRB Protocol #H18-220, #H15-183, and #H10-043).

Pre-Testing Procedures The initial Climatic Chamber Testing Session can be completed after approximately 48 hours have passed since the completion of all Session 1 baseline testing procedures. This time period would include the completion of both the phase specific Baseline Visit and Dehydration Period. Phases 2, 3, 4, and 5 will be completed approximately 24 hours the completion of their phase specific Baseline Visit where participants will be instructed to arrive at the HPL at the cessation of their Dehydration Period. Similar to Session 1, participants will be instructed to refrain from eating or smoking for up to 3 hours before the beginning of their testing session. Additionally, participants will be instructed to partake in an 18-24-hour fluid restriction period in order to exacerbate the dehydrated response to both passive and exertional heat stress. For testing sessions only, upon arrival participants will be asked to complete a nude body mass in private to confirm that they have achieved the desired level of dehydration from their baseline (~1.5-3%). In addition to the body mass loss, participants will also be asked to provide their 24-hour urine sample (collected during the dehydration period) and a spot urine sample. The spot urine sample will be used to confirm dehydration indicated by a USG >1.024, however this urinary measure will not exclude participation but rather confirm the participant's hydration status. Next, the participant will be asked to don a heart rate strap and provide their completed thirst scale and dietary recall log. Upon completion, resting cardiovascular measurements will be collected including HRV, HR, and BP. Once completed, the participant will complete the cognitive/performance battery which will include completion of the ANAM testing battery, BESS, and hand grip strength and endurance. Afterwards, participants will have a venous cannula inserted by an HPL trained research team member to allow for subsequent sampling of blood without the need for multiple needle sticks. Upon a successful insertion of the venous cannula a blood draw will be completed for the collection of 11 mL (~0.75 tablespoon) of blood. Afterwards, the participant will have the Nix Biosensor applied to the pre-determined location on their body (between the belly button and the rib cage) and will be provided the predetermined amount (i.e., 0.8g/kg or 0.4g/kg) of the biomedical intervention supplement (i.e., PR or Placebo Lotion) to be applied to their entire body (from neck to ankles) within the privacy of a restroom. Finally, prior to entering the environmental chamber, participants will be instructed to privately insert the rectal thermometer 10-15 cm beyond the anal sphincter for the continuous monitoring of core body temperature.

Data Collection - Initial 95 minutes Once the subject has indicated they have successfully completed all required arrival procedures, they will then be permitted to enter the environmental chamber (~330C [91.40F], ~25% relative humidity) where they will be instructed to sit down at a desk provided and begin a 15-minute period of environmental equilibration. At the end of the environmental equilibration, identified as time point 0 in Figure 7, the participant will be asked to complete an HRV assessment before having another 11mL blood sample, nude body mass, and spot urine sample collected. Similar assessments will be completed at time point 40. At time point 80, similar assessments will be completed in addition to the cognitive battery (ANAM testing battery) and the performance battery (BESS and hand grip strength and endurance). Furthermore, 2 additional 3 mL blood samples (~1 teaspoon total) will be collected at time points 20 and 60 of the protocol as illustrated in Figure 7. Finally, three equal fluid boluses will be provided for three of the proposed phases to be completed (0.8PR - Fluid, 0.4PR - Fluid, PLA - Fluid) at the 10-, 20-, and 30- minute marks as illustrated in Figure 7. The fluid bolus amount will be relative to the subject's body composition and will be enough to replace ~1% of the body mass lost between body mass measured on the intervention trial day and body mass measured during their initial baseline visit (Session 1). This fluid bolus will be provided for the assessment of fluid retention in regards to the biomedical intervention and its associated amount applied to the participant's body.

Data Collection - 120-minute Exercise Protocol At the completion of all data collection procedures conducted at the 80-minute mark (i.e., passive heat stress), the participant will immediately be escorted to the treadmill for the initiation of their exercise protocol. The protocol will include the completion of aerobic exercise (walking or jogging) conducted at ~40% of the participant's velocity measured during the last stage of their baseline VO2max test (i.e., vVO2max). This portion of the protocol (i.e., exertional heat stress) will begin with the participant donning the Hans Rudolph mask which will be attached to a breathing tube for the measurement of expired air delivered to the metabolic cart system during the exercise protocol. Similar to measurements collected during the participant's baseline VO2max test, the metabolic cart will continuously measure respiratory exchange ratio (RER), oxygen consumption (VO2), and carbon dioxide production (VCO2) while being used by the participant. This assessment will be used during three separate 5-minute intervals at the 100-, 160-, and 215-minute marks. Aerobic exercise completed between these time points will not require the subject to wear the Hans Rudolph mask as indicated in Figure 7. Using the previously inserted cannula, supplemental 3 mL blood draws will be completed at the 130- and 190-minute marks. Additionally, one 11 mL blood draw will be completed at the 220-minute time mark. Finally, assessments will be completed immediately after the completion of the exercise protocol and will include the assessment of the participant's nude body mass and collection of a spot urine sample in addition to assessment of the participants cardiovascular health (i.e., HR, HRV, and BP) and completion of the cognitive battery (ANAM testing battery) and performance tasks (BESS, hand grip strength, and hand grip endurance). Once all measurements have been collected the participant will be directed to exit the environmental chamber for the completion of their discharge from the HPL.

Sub-study - 24-hour Rehydration Sessions At the completion of the participant's discharge procedures, the participant will initiate their 24-hour recovery period where the progression of their rehydration during the post-exercise recovery period will be compared between the provision of one of two amino acid rehydration beverages (i.e., AminoVITAL Rapid Recovery or Placebo). For the completion of comparisons between these two beverages, participants will be matched on demographical information pertaining to their aerobic fitness level (i.e., VO2max), body mass index (BMI), body surface area (BSA), and/or age. Once identified, the beverage will be provided to the participant before the completion of each of their discharge protocols to ensure completion for the 24-hour follow-up session. Moreover, participants will be provided specific instructions pertaining to consistency in regards to their nutritional intake and fluid consumption over the 24-hour period following exercise until they are directed to come back to the HPL for the completion of follow-up testing procedures.

Rehydration Protocol Before departing the HPL, participants will be provided four separate bags where each will include all of the following items: (1) one jug provided for the collection of urine throughout the predetermined time period; (2) one urine cup for the collection of a spot urine sample at the end of each predetermined time period; (3) two perceptual questionnaires (i.e., AD-ACL and CFS) for completion at the end of each predetermined time period; and (4) the predetermined nutritional supplement (AminoVITAL Rapid Recovery or Placebo) to be consumed at the beginning of each predetermined time period (See illustration of timeline in Figure 8). Participants will be instructed on storage of all materials and will be required to return all completed materials and collected biospecimens upon their return to the HPL approximately 24-hours after the completion of their testing session.

Topical Solution Procedures Supplies containing the topical solution will be provided to the participant for application to their body within the privacy of a restroom. The amount of lotion provided for application will be dependent on the session completed (i.e., 0.8g/kg or 0.4g/kg) and relative to the participant's body composition. To ensure the product usage adheres to the drug facts label provided, research team personnel will ensure that the bottle is well shaken prior to dispensing the lotion into the plastic bag. When it is time to apply the product to their body, the participant will be instructed to wash their hands before and after applying the product in addition to avoiding contact with any open orifices on their face (i.e., eyes, mouth, nose, etc.) until their hands have been washed. In efforts to keep the lotion from the participant's hands, the lotion will be provided within a plastic bag and the participant will be instructed to insert their hand into the opposite side of the bag while directly applying the lotion to the body from the bag. After the lotion has been appropriately applied, the participant will return the used bag to the research team member so that pre-application and post-application weight can be measured and compared for proper assessment of lotion amount applied to the skin. Participants will be instructed to apply the solution primarily to areas of their lower extremities (i.e., thighs, hamstrings, calves, buttocks, etc.) in addition to their lower back, arms, midsection, and/or chest if enough solution is available. Application will be considered complete when the solution has been transmitted to the skin in a fashion where no residue from the lotion is visible by researchers from the skin of the participant.

Collection of Urine Samples and Body Weight Measurements For the collection of all urine spot samples, researchers will provide a clean cup and top to seal the capsule. Participants will be asked to provide a sample regardless of urgency to urinate at specific time points during the trial. If the participant is unable to provide a sample at the time point requested, no protocol deviation will be considered as the lack in sample provided will still be used towards the completion of data analysis. Furthermore, if the participant must provide a urine sample without being requested by a research team member, any urine expelled will be added to the amount collected (if any) during the next urine sample collection time point. Additionally, participants will be instructed to complete a measurement of nude body weight completed before the provision of a urine sample. Both the collection of urine samples and measurement of body weight will be completed within the privacy of a bathroom.

ELIGIBILITY:
Inclusion Criteria:

1. Males within the age range of 18- 45 years old.
2. Individuals who are classified as recreationally active adults as indicated by a VO2max minimum (45 ml/kg/min)
3. Individuals who measure with a BMI of ≤ 28
4. Individuals who have been medically cleared for participation in this study by the medical safety monitor.

Exclusion Criteria:

1. Cannot understand English (written and/or verbally communicated).
2. Hearing impaired to where verbal communications cannot be understood and/or followed safely.
3. Individuals who report a history of COVID-19 unless cleared by a physician for exercise at the performance level required to participate in this study. The physician must be made aware of what is required to participate in this study.
4. Individuals who self-report history of complications with psychological disorders or chronic illness (eating disorders, cardiovascular, kidney, liver, metabolic, neuromuscular, pulmonary, integumentary, and/or sickle cell disease).
5. Individuals who have chronic health problems that may affect the participant's ability to thermoregulate or sweat normally.
6. Individuals who have a history of exertional heat illness within the past 3 years.
7. Individuals who are taking any prescription or non-prescription medication(s) that may specifically impact cardiometabolic, pulmonary, renal, integumentary, and/or thermoregulatory function (i.e. amphetamines, antihypertensives, anticholinergics, acetaminophen, NSAIDs, aspirin, and water pills).
8. Individuals who are taking any prescription medication for diabetes mellitus, Parkinson's disease, or kidney disease.
9. Individuals who have donated blood within the previous month.
10. Individuals who have an implanted pacemaker or internal defibrillator.
11. Individuals who report a history of claustrophobia
12. Individuals classified as hypertensive while at rest (SBP: ≥140 mmHg and/or DBP: ≥90 mmHg; will be measured during first visit).
13. Individuals who have not abstained from use of supplements that may affect/enhance hydration status and/or rehydration protocol measurements (i.e. creatine, sodium bicarbonate, potassium, magnesium, dandelion, vitamin B, protein powder, BCAAs, fish oil, multivitamins, soluble fiber, other natural diuretics) at time of testing.
14. Individuals who are suffering from a current musculoskeletal injury or active lesion of the skin that inhibits the participant's ability to complete all tasks required for participation.
15. Individuals who are allergic/sensitive to adhesive materials (i.e., medical tape)
16. Individuals who are allergic/sensitive to ingredients within the study-specific Topical Lotions: (Menthol [0.5%], sodium bicarbonate (baking soda), water, isopropyl palmitate, lecithin, poloxamer 407, cetyl alcohol, propylene glycol, denatured alcohol, benzyl alcohol, polyglyceryl-4 laurate, sodium hydroxide, sodium lauryl sulfate, sorbic acid, and fragrance) as well as iodine and/or medical tape.
17. Individuals who are allergic/sensitive to ingredients within the study specific amino acid beverages: highly branched cyclic dextrin, citric acid, malic acid, natural fruit flavor, rebaudioside (stevia leaf extract), and vegetable juice for color.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Hydration Status - Change in Acute Urine USG | Phase-specific PRE Session
  Assessment of hydration status via collection of urine USG
Hydration Status - Change in 24-h Urine USG | Phase-specific PRE Session
  Assessment of hydration status via collection of urine USG
Hydration Status - Change in Acute Urine USG | Intervention Trial at the -45 minute mark
  Assessment of hydration status via collection of urine USG
Hydration Status - Change in 24-h Urine USG | Intervention Trial at the -45 minute mark
  Assessment of hydration status via collection of urine USG
Hydration Status - Change in Urine USG | Intervention Trial at the 0 minute mark
  Assessment of hydration status via collection of urine USG
Hydration Status - Change in Urine USG | Intervention Trial at the 40 minute mark
  Assessment of hydration status via collection of urine USG
Hydration Status - Change in Acute Urine USG | Intervention Trial at the 80 minute mark
  Assessment of hydration status via collection of urine USG
Hydration Status - Change in Urine USG | Intervention Trial at the 220 minute mark
  Assessment of hydration status via collection of urine USG
Hydration Status - Change in Urine USG | Rehydration Protocol - 3 hours post-intervention
  Assessment of hydration status via collection of urine USG
Hydration Status - Change in Urine USG | Rehydration Protocol - 6 hours post-intervention
  Assessment of hydration status via collection of urine USG
Hydration Status - Change in Urine USG | Rehydration Protocol -15 hours post-intervention
  Assessment of hydration status via collection of urine USG
Hydration Status - Change in Urine USG | Rehydration Protocol - 24 hours post-intervention
  Assessment of hydration status via collection of urine USG
Hydration Status - Change in Acute Urine Osmolality | Phase-specific PRE Session
  Assessment of hydration status via collection of urine osmolality
Hydration Status - Change in 24-h Urine Osmolality | Phase-specific PRE Session
  Assessment of hydration status via collection of urine osmolality
Hydration Status - Change in Acute Urine Osmolality | Intervention Trial at the -45 minute mark
  Assessment of hydration status via collection of urine osmolality
Hydration Status - Change in 24-h Urine Osmolality | Intervention Trial at the -45 minute mark
  Assessment of hydration status via collection of urine osmolality
Hydration Status - Change in Urine Osmolality | Intervention Trial at the 0 minute mark
  Assessment of hydration status via collection of urine osmolality
Hydration Status - Change in Urine Osmolality | Intervention Trial at the 40 minute mark
  Assessment of hydration status via collection of urine osmolality
Hydration Status - Change in Urine Osmolality | Intervention Trial at the 80 minute mark
  Assessment of hydration status via collection of urine osmolality
Hydration Status - Change in Urine Osmolality | Intervention Trial at the 220 minute mark
  Assessment of hydration status via collection of urine osmolality
Hydration Status - Change in Urine Osmolality | Rehydration Protocol - 3 hours post-intervention
  Assessment of hydration status via collection of urine osmolality
Hydration Status - Change in Urine Osmolality | Rehydration Protocol - 6 hours post-intervention
  Assessment of hydration status via collection of urine osmolality
Hydration Status - Change in Urine Osmolality | Rehydration Protocol - 15 hours post-intervention
  Assessment of hydration status via collection of urine osmolality
Hydration Status - Change in Urine Osmolality | Rehydration Protocol - 24 hours post-intervention
  Assessment of hydration status via collection of urine osmolality
Renal Electrolyte Levels - Change in Acute Urine Sodium | Phase-specific PRE Session
  Assessment of renal electrolyte levels via collection of urine sodium excretion
Renal Electrolyte Levels - Change in 24-h Urine Sodium | Phase-specific PRE Session
  Assessment of renal electrolyte levels via collection of urine sodium excretion
Renal Electrolyte Levels - Change in Acute Urine Sodium | Intervention Trial at the -45 minute mark
  Assessment of renal electrolyte levels via collection of urine sodium excretion
Renal Electrolyte Levels - Change in 24-h Urine Sodium | Intervention Trial at the -45 minute mark
  Assessment of renal electrolyte levels via collection of urine sodium excretion
Renal Electrolyte Levels - Change in Urine Sodium | Intervention Trial at the 0 minute mark
  Assessment of renal electrolyte levels via collection of urine sodium excretion
Renal Electrolyte Levels - Change in Urine Sodium | Intervention Trial at the 40 minute mark
  Assessment of renal electrolyte levels via collection of urine sodium excretion
Renal Electrolyte Levels - Change in Urine Sodium | Intervention Trial at the 80 minute mark
  Assessment of renal electrolyte levels via collection of urine sodium excretion
Renal Electrolyte Levels - Change in Urine Sodium | Intervention Trial at the 220 minute mark
  Assessment of renal electrolyte levels via collection of urine sodium excretion
Renal Electrolyte Levels - Change in Urine Sodium | Rehydration Protocol - 3 hours post-intervention
  Assessment of renal electrolyte levels via collection of urine sodium excretion
Renal Electrolyte Levels - Change in Urine Sodium | Rehydration Protocol - 6 hours post-intervention
  Assessment of renal electrolyte levels via collection of urine sodium excretion
Renal Electrolyte Levels - Change in Urine Sodium | Rehydration Protocol - 15 hours post-intervention
  Assessment of renal electrolyte levels via collection of urine sodium excretion
Renal Electrolyte Levels - Change in Urine Sodium | Rehydration Protocol - 24 hours post-intervention
  Assessment of renal electrolyte levels via collection of urine sodium excretion
Renal Electrolyte Levels - Change in Acute Urine Potassium | Phase-specific PRE Session
  Assessment of renal electrolyte levels via collection of urine potassium excretion
Renal Electrolyte Levels - Change in 24-h Urine Potassium | Phase-specific PRE Session
  Assessment of renal electrolyte levels via collection of urine potassium excretion
Renal Electrolyte Levels - Change in Acute Urine Potassium | Intervention Trial at the -45 minute mark
  Assessment of renal electrolyte levels via collection of urine potassium excretion
Renal Electrolyte Levels - Change in 24-h Urine Potassium | Intervention Trial at the -45 minute mark
  Assessment of renal electrolyte levels via collection of urine potassium excretion
Renal Electrolyte Levels - Change in Urine Potassium | Intervention Trial at the 0 minute mark
  Assessment of renal electrolyte levels via collection of urine potassium excretion
Renal Electrolyte Levels - Change in Urine Potassium | Intervention Trial at the 40 minute mark
  Assessment of renal electrolyte levels via collection of urine potassium excretion
Renal Electrolyte Levels - Change in Urine Potassium | Intervention Trial at the 80 minute mark
  Assessment of renal electrolyte levels via collection of urine potassium excretion
Renal Electrolyte Levels - Change in Urine Potassium | Intervention Trial at the 220 minute mark
  Assessment of renal electrolyte levels via collection of urine potassium excretion
Renal Electrolyte Levels - Change in Urine Potassium | Rehydration Protocol - 3 hours post-intervention
  Assessment of renal electrolyte levels via collection of urine potassium excretion
Renal Electrolyte Levels - Change in Urine Potassium | Rehydration Protocol - 6 hours post-intervention
  Assessment of renal electrolyte levels via collection of urine potassium excretion
Renal Electrolyte Levels - Change in Urine Potassium | Rehydration Protocol - 15 hours post-intervention
  Assessment of renal electrolyte levels via collection of urine potassium excretion
Renal Electrolyte Levels - Change in Urine Potassium | Rehydration Protocol - 24 hours post-intervention
  Assessment of renal electrolyte levels via collection of urine potassium excretion
Renal Electrolyte Levels - Change in Acute Urine Chloride | Phase-specific PRE Session
  Assessment of renal electrolyte levels via collection of urine chloride excretion
Renal Electrolyte Levels - Change in 24-h Urine Chloride | Phase-specific PRE Session
  Assessment of renal electrolyte levels via collection of urine chloride excretion
Renal Electrolyte Levels - Change in Acute Urine Chloride | Intervention Trial at the -45 minute mark
  Assessment of renal electrolyte levels via collection of urine chloride excretion
Renal Electrolyte Levels - Change in 24-h Urine Chloride | Intervention Trial at the -45 minute mark
  Assessment of renal electrolyte levels via collection of urine chloride excretion
Renal Electrolyte Levels - Change in Urine Chloride | Intervention Trial at the 0 minute mark
  Assessment of renal electrolyte levels via collection of urine chloride excretion
Renal Electrolyte Levels - Change in Urine Chloride | Intervention Trial at the 40 minute mark
  Assessment of renal electrolyte levels via collection of urine chloride excretion
Renal Electrolyte Levels - Change in Urine Chloride | Intervention Trial at the 80 minute mark
  Assessment of renal electrolyte levels via collection of urine chloride excretion
Renal Electrolyte Levels - Change in Urine Chloride | Intervention Trial at the 220 minute mark
  Assessment of renal electrolyte levels via collection of urine chloride excretion
Renal Electrolyte Levels - Change in Urine Chloride | Rehydration Protocol - 3 hours post-intervention
  Assessment of renal electrolyte levels via collection of urine chloride excretion
Renal Electrolyte Levels - Change in Urine Chloride | Rehydration Protocol - 6 hours post-intervention
  Assessment of renal electrolyte levels via collection of urine chloride excretion
Renal Electrolyte Levels - Change in Urine Chloride | Rehydration Protocol - 15 hours post-intervention
  Assessment of renal electrolyte levels via collection of urine chloride excretion
Renal Electrolyte Levels - Change in Urine Chloride | Rehydration Protocol - 24 hours post-intervention
  Assessment of renal electrolyte levels via collection of urine chloride excretion
Systemic Electrolyte Levels - Change in Plasma Sodium | Phase-specific PRE Session
  Assessment of circulatory electrolyte levels via collection of plasma sodium levels
Systemic Electrolyte Levels - Change in Plasma Sodium | Intervention Trial at the -35 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma sodium levels
Systemic Electrolyte Levels - Change in Plasma Sodium | Intervention Trial at the 0 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma sodium levels
Systemic Electrolyte Levels - Change in Plasma Sodium | Intervention Trial at the 20 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma sodium levels
Systemic Electrolyte Levels - Change in Plasma Sodium | Intervention Trial at the 40 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma sodium levels
Systemic Electrolyte Levels - Change in Plasma Sodium | Intervention Trial at the 60 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma sodium levels
Systemic Electrolyte Levels - Change in Plasma Sodium | Intervention Trial at the 80 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma sodium levels
Systemic Electrolyte Levels - Change in Plasma Sodium | Intervention Trial at the 130 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma sodium levels
Systemic Electrolyte Levels - Change in Plasma Sodium | Intervention Trial at the 190 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma sodium levels
Systemic Electrolyte Levels - Change in Plasma Sodium | Intervention Trial at the 220 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma sodium levels
Systemic Electrolyte Levels - Change in Plasma Sodium | Rehydration Protocol - 24 hours post-intervention
  Assessment of circulatory electrolyte levels via collection of plasma sodium levels
Systemic Electrolyte Levels - Change in Plasma Potassium | Phase-specific PRE Session
  Assessment of circulatory electrolyte levels via collection of plasma potassium levels
Systemic Electrolyte Levels - Change in Plasma Potassium | Intervention Trial at the -35 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma potassium levels
Systemic Electrolyte Levels - Change in Plasma Potassium | Intervention Trial at the 0 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma potassium levels
Systemic Electrolyte Levels - Change in Plasma Potassium | Intervention Trial at the 20 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma potassium levels
Systemic Electrolyte Levels - Change in Plasma Potassium | Intervention Trial at the 40 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma potassium levels
Systemic Electrolyte Levels - Change in Plasma Potassium | Intervention Trial at the 60 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma potassium levels
Systemic Electrolyte Levels - Change in Plasma Potassium | Intervention Trial at the 80 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma potassium levels
Systemic Electrolyte Levels - Change in Plasma Potassium | Intervention Trial at the 220 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma potassium levels
Systemic Electrolyte Levels - Change in Plasma Potassium | Rehydration Protocol - 24 hours post-intervention
  Assessment of circulatory electrolyte levels via collection of plasma potassium levels
Systemic Electrolyte Levels - Change in Plasma Chloride | Phase-specific PRE Session
  Assessment of circulatory electrolyte levels via collection of plasma chloride levels
Systemic Electrolyte Levels - Change in Plasma Chloride | Intervention Trial at the -35 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma chloride levels
Systemic Electrolyte Levels - Change in Plasma Chloride | Intervention Trial at the 0 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma chloride levels
Systemic Electrolyte Levels - Change in Plasma Chloride | Intervention Trial at the 20 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma chloride levels
Systemic Electrolyte Levels - Change in Plasma Chloride | Intervention Trial at the 40 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma chloride levels
Systemic Electrolyte Levels - Change in Plasma Chloride | Intervention Trial at the 60 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma chloride levels
Systemic Electrolyte Levels - Change in Plasma Chloride | Intervention Trial at the 80 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma chloride levels
Systemic Electrolyte Levels - Change in Plasma Chloride | Intervention Trial at the 130 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma chloride levels
Systemic Electrolyte Levels - Change in Plasma Chloride | Intervention Trial at the 190 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma chloride levels
Systemic Electrolyte Levels - Change in Plasma Chloride | Intervention Trial at the 220 minute mark
  Assessment of circulatory electrolyte levels via collection of plasma chloride levels
Systemic Electrolyte Levels - Change in Plasma Chloride | Rehydration Protocol - 24 hours post-intervention
  Assessment of circulatory electrolyte levels via collection of plasma chloride levels
Systemic Osmotic Stress - Change in Plasma Osmolality | Phase-specific PRE Session
  Assessment of circulatory osmotic stress levels via collection of plasma osmolality levels
Systemic Osmotic Stress - Change in Plasma Osmolality | Intervention Trial at the -35 minute mark
  Assessment of circulatory osmotic stress levels via collection of plasma osmolality levels
Systemic Osmotic Stress - Change in Plasma Osmolality | Intervention Trial at the 0 minute mark
  Assessment of circulatory osmotic stress levels via collection of plasma osmolality levels
Systemic Osmotic Stress - Change in Plasma Osmolality | Intervention Trial at the 20 minute mark
  Assessment of circulatory osmotic stress levels via collection of plasma osmolality levels
Systemic Osmotic Stress - Change in Plasma Osmolality | Intervention Trial at the 40 minute mark
  Assessment of circulatory osmotic stress levels via collection of plasma osmolality levels
Systemic Osmotic Stress - Change in Plasma Osmolality | Intervention Trial at the 60 minute mark
  Assessment of circulatory osmotic stress levels via collection of plasma osmolality levels
Systemic Osmotic Stress - Change in Plasma Osmolality | Intervention Trial at the 80 minute mark
  Assessment of circulatory osmotic stress levels via collection of plasma osmolality levels
Systemic Osmotic Stress - Change in Plasma Osmolality | Intervention Trial at the 130 minute mark
  Assessment of circulatory osmotic stress levels via collection of plasma osmolality levels
Systemic Osmotic Stress - Change in Plasma Osmolality | Intervention Trial at the 190 minute mark
  Assessment of circulatory osmotic stress levels via collection of plasma osmolality levels
Systemic Osmotic Stress - Change in Plasma Osmolality | Intervention Trial at the 220 minute mark
  Assessment of circulatory osmotic stress levels via collection of plasma osmolality levels
Systemic Osmotic Stress - Change in Plasma Osmolality | Rehydration Protocol - 24 hours post-intervention
  Assessment of circulatory osmotic stress levels via collection of plasma osmolality levels
Renal Function - Change in Acute Urinary Creatinine Levels | Phase-specific PRE Session
  Assessment of renal function and potential sustainment of injury via collection of urinary creatinine levels
Renal Function - Change in 24-h Urinary Creatinine Levels | Phase-specific PRE Session
  Assessment of renal function and potential sustainment of injury via collection of urinary creatinine levels
Renal Function - Change in Acute Urinary Creatinine Levels | Intervention Trial at the -45 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary creatinine levels
Renal Function - Change in Acute Urinary Creatinine Levels | Intervention Trial at the 0 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary creatinine levels
Renal Function - Change in Acute Urinary Creatinine Levels | Intervention Trial at the 40 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary creatinine levels
Renal Function - Change in Acute Urinary Creatinine Levels | Intervention Trial at the 80 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary creatinine levels
Renal Function - Change in Acute Urinary Creatinine Levels | Intervention Trial at the 220 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary creatinine levels
Renal Function - Change in Urinary Creatinine Levels | Rehydration Protocol - 3 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary creatinine levels
Renal Function - Change in Urinary Creatinine Levels | Rehydration Protocol - 6 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary creatinine levels
Renal Function - Change in Urinary Creatinine Levels | Rehydration Protocol - 15 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary creatinine levels
Renal Function - Change in Urinary Creatinine Levels | Rehydration Protocol - 24 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary creatinine levels
Renal Function - Change in Acute Urinary BUN Levels | Phase-specific PRE Session
  Assessment of renal function and potential sustainment of injury via collection of urinary BUN levels
Renal Function - Change in 24-h Urinary BUN Levels | Phase-specific PRE Session
  Assessment of renal function and potential sustainment of injury via collection of urinary BUN levels
Renal Function - Change in Acute Urinary BUN Levels | Intervention Trial at the -45 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary BUN levels
Renal Function - Change in Chronic Urinary BUN Levels | Intervention Trial at the -45 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary BUN levels
Renal Function - Change in Urinary BUN Levels | Intervention Trial at the 0 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary BUN levels
Renal Function - Change in Urinary BUN Levels | Intervention Trial at the 40 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary BUN levels
Renal Function - Change in Urinary BUN Levels | Intervention Trial at the 80 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary BUN levels
Renal Function - Change in Urinary BUN Levels | Intervention Trial at the 220 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary BUN levels
Renal Function - Change in Urinary BUN Levels | Rehydration Protocol - 3 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary BUN levels
Renal Function - Change in Urinary BUN Levels | Rehydration Protocol - 6 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary BUN levels
Renal Function - Change in Urinary BUN Levels | Rehydration Protocol - 15 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary BUN levels
Renal Function - Change in Urinary BUN Levels | Rehydration Protocol - 24 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary BUN levels
Renal Function - Change in Acute Urinary IGFBP7 Levels | Phase-specific PRE Session
  Assessment of renal function and potential sustainment of injury via collection of urinary IGFBP7 levels
Renal Function - Change in 24-h Urinary IGFBP7 Levels | Phase-specific PRE Session
  Assessment of renal function and potential sustainment of injury via collection of urinary IGFBP7 levels
Renal Function - Change in Acute Urinary IGFBP7 Levels | Intervention Trial at the -45 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary IGFBP7 levels
Renal Function - Change in 24-h Urinary IGFBP7 Levels | Intervention Trial at the -45 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary IGFBP7 levels
Renal Function - Change in Urinary IGFBP7 Levels | Intervention Trial at the 0 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary IGFBP7 levels
Renal Function - Change in Urinary IGFBP7 Levels | Intervention Trial at the 40 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary IGFBP7 levels
Renal Function - Change in Urinary IGFBP7 Levels | Intervention Trial at the 80 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary IGFBP7 levels
Renal Function - Change in Urinary IGFBP7 Levels | Intervention Trial at the 220 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary IGFBP7 levels
Renal Function - Change in Urinary IGFBP7 Levels | Rehydration Protocol - 3 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary IGFBP7 levels
Renal Function - Change in Urinary IGFBP7 Levels | Rehydration Protocol - 6 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary IGFBP7 levels
Renal Function - Change in Urinary IGFBP7 Levels | Rehydration Protocol - 15 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary IGFBP7 levels
Renal Function - Change in Urinary IGFBP7 Levels | Rehydration Protocol - 24 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary IGFBP7 levels
Renal Function - Change in Acute Urinary TIMP2 Levels | Phase-specific PRE Session
  Assessment of renal function and potential sustainment of injury via collection of urinary TIMP2 levels
Renal Function - Change in 24-h Urinary TIMP2 Levels | Phase-specific PRE Session
  Assessment of renal function and potential sustainment of injury via collection of urinary TIMP2 levels
Renal Function - Change in Acute Urinary TIMP2 Levels | Intervention Trial at the -45 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary TIMP2 levels
Renal Function - Change in 24-h Urinary TIMP2 Levels | Intervention Trial at the -45 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary TIMP2 levels
Renal Function - Change in Urinary TIMP2 Levels | Intervention Trial at the 0 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary TIMP2 levels
Renal Function - Change in Urinary TIMP2 Levels | Intervention Trial at the 40 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary TIMP2 levels
Renal Function - Change in Urinary TIMP2 Levels | Intervention Trial at the 80 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary TIMP2 levels
Renal Function - Change in Urinary TIMP2 Levels | Intervention Trial at the 220 minute mark
  Assessment of renal function and potential sustainment of injury via collection of urinary TIMP2 levels
Renal Function - Change in Urinary TIMP2 Levels | Rehydration Protocol - 3 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary TIMP2 levels
Renal Function - Change in Urinary TIMP2 Levels | Rehydration Protocol - 6 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary TIMP2 levels
Renal Function - Change in Urinary TIMP2 Levels | Rehydration Protocol - 15 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary TIMP2 levels
Renal Function - Change in Urinary TIMP2 Levels | Rehydration Protocol - 24 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of urinary TIMP2 levels
Renal Function - Change in Plasma Creatinine Levels | Phase-specific PRE Session
  Assessment of renal function and potential sustainment of injury via collection of plasma creatinine levels
Renal Function - Change in Plasma Creatinine Levels | Intervention Trial at the -35 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma creatinine levels
Renal Function - Change in Plasma Creatinine Levels | Intervention Trial at the 0 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma creatinine levels
Renal Function - Change in Plasma Creatinine Levels | Intervention Trial at the 40 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma creatinine levels
Renal Function - Change in Plasma Creatinine Levels | Intervention Trial at the 80 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma creatinine levels
Renal Function - Change in Plasma Creatinine Levels | Intervention Trial at the 220 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma creatinine levels
Renal Function - Change in Plasma Creatinine Levels | Rehydration Protocol - 24 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of plasma creatinine levels
Renal Function - Change in Plasma BUN Levels | Phase-specific PRE Session
  Assessment of renal function and potential sustainment of injury via collection of plasma BUN levels
Renal Function - Change in Plasma BUN Levels | Intervention Trial at the -35 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma BUN levels
Renal Function - Change in Plasma BUN Levels | Intervention Trial at the 0 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma BUN levels
Renal Function - Change in Plasma BUN Levels | Intervention Trial at the 40 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma BUN levels
Renal Function - Change in Plasma BUN Levels | Intervention Trial at the 80 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma BUN levels
Renal Function - Change in Plasma BUN Levels | Intervention Trial at the 220 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma BUN levels
Renal Function - Change in Plasma BUN Levels | Rehydration Protocol - 24 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of plasma BUN levels
Renal Function - Change in Plasma IGFBP7 Levels | Phase-specific PRE Session
  Assessment of renal function and potential sustainment of injury via collection of plasma IGFBP7 levels
Renal Function - Change in Plasma IGFBP7 Levels | Intervention Trial at -35 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma IGFBP7 levels
Renal Function - Change in Plasma IGFBP7 Levels | Intervention Trial at 0 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma IGFBP7 levels
Renal Function - Change in Plasma IGFBP7 Levels | Intervention Trial at 40 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma IGFBP7 levels
Renal Function - Change in Plasma IGFBP7 Levels | Intervention Trial at 80 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma IGFBP7 levels
Renal Function - Change in Plasma IGFBP7 Levels | Intervention Trial at 220 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma IGFBP7 levels
Renal Function - Change in Plasma IGFBP7 Levels | Rehydration Protocol - 24 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of plasma IGFBP7 levels
Renal Function - Change in Plasma TIMP2 Levels | Phase-specific PRE Session
  Assessment of renal function and potential sustainment of injury via collection of plasma TIMP2 levels
Renal Function - Change in Plasma TIMP2 Levels | Intervention Trial at the -35 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma TIMP2 levels
Renal Function - Change in Plasma TIMP2 Levels | Intervention Trial at the 0 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma TIMP2 levels
Renal Function - Change in Plasma TIMP2 Levels | Intervention Trial at the 40 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma TIMP2 levels
Renal Function - Change in Plasma TIMP2 Levels | Intervention Trial at the 80 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma TIMP2 levels
Renal Function - Change in Plasma TIMP2 Levels | Intervention Trial at the 220 minute mark
  Assessment of renal function and potential sustainment of injury via collection of plasma TIMP2 levels
Renal Function - Change in Plasma TIMP2 Levels | Rehydration Protocol - 24 hours post-intervention
  Assessment of renal function and potential sustainment of injury via collection of plasma TIMP2 levels

SECONDARY OUTCOMES:
Hydration Status - Change in Whole Blood Plasma Volume Shifts | Phase-specific PRE Session
  Assessment of whole blood hematocrit and hemoglobin for evaluation of acute plasma volume shifts within biological sample collected reported as a percentage (%)
Hydration Status - Change in Whole Blood Plasma Volume Shifts | Intervention Trial at the -35 minute mark
  Assessment of whole blood hematocrit and hemoglobin for evaluation of acute plasma volume shifts within biological sample collected reported as a percentage (%)
Hydration Status - Change in Whole Blood Plasma Volume Shifts | Intervention Trial at the 0 minute mark
  Assessment of whole blood hematocrit and hemoglobin for evaluation of acute plasma volume shifts within biological sample collected reported as a percentage (%)
Hydration Status - Change in Whole Blood Plasma Volume Shifts | Intervention Trial at the 20 minute mark
  Assessment of whole blood hematocrit and hemoglobin for evaluation of acute plasma volume shifts within biological sample collected reported as a percentage (%)
Hydration Status - Change in Whole Blood Plasma Volume Shifts | Intervention Trial at the 40 minute mark
  Assessment of whole blood hematocrit and hemoglobin for evaluation of acute plasma volume shifts within biological sample collected reported as a percentage (%)
Hydration Status - Change in Whole Blood Plasma Volume Shifts | Intervention Trial at the 60 minute mark
  Assessment of whole blood hematocrit and hemoglobin for evaluation of acute plasma volume shifts within biological sample collected reported as a percentage (%)
Hydration Status - Change in Whole Blood Plasma Volume Shifts | Intervention Trial at the 80 minute mark
  Assessment of whole blood hematocrit and hemoglobin for evaluation of acute plasma volume shifts within biological sample collected reported as a percentage (%)
Hydration Status - Change in Whole Blood Plasma Volume Shifts | Intervention Trial at the 130 minute mark
  Assessment of whole blood hematocrit and hemoglobin for evaluation of acute plasma volume shifts within biological sample collected reported as a percentage (%)
Hydration Status - Change in Whole Blood Plasma Volume Shifts | Intervention Trial at the 190 minute mark
  Assessment of whole blood hematocrit and hemoglobin for evaluation of acute plasma volume shifts within biological sample collected reported as a percentage (%)
Hydration Status - Change in Whole Blood Plasma Volume Shifts | Intervention Trial at the 220 minute mark
  Assessment of whole blood hematocrit and hemoglobin for evaluation of acute plasma volume shifts within biological sample collected reported as a percentage (%)
Hydration Status - Change in Whole Blood Plasma Volume Shifts | Rehydration Protocol - 24 hours post-intervention
  Assessment of whole blood hematocrit and hemoglobin for evaluation of acute plasma volume shifts within biological sample collected reported as a percentage (%)
Protein Content - Change in Plasma Protein Levels | Phase-specific PRE Session
  Assessment of plasma protein levels within biospecimen samples collected.
Protein Content - Change in Plasma Protein Levels | Intervention Trial at the -35 minute mark
  Assessment of plasma protein levels within biospecimen samples collected.
Protein Content - Change in Plasma Protein Levels | Intervention Trial at the 0 minute mark
  Assessment of plasma protein levels within biospecimen samples collected.
Protein Content - Change in Plasma Protein Levels | Intervention Trial at the 20 minute mark
  Assessment of plasma protein levels within biospecimen samples collected.
Protein Content - Change in Plasma Protein Levels | Intervention Trial at the 40 minute mark
  Assessment of plasma protein levels within biospecimen samples collected.
Protein Content - Change in Plasma Protein Levels | Intervention Trial at the 60 minute mark
  Assessment of plasma protein levels within biospecimen samples collected.
Protein Content - Change in Plasma Protein Levels | Intervention Trial at the 80 minute mark
  Assessment of plasma protein levels within biospecimen samples collected.
Protein Content - Change in Plasma Protein Levels | Intervention Trial at the 130 minute mark
  Assessment of plasma protein levels within biospecimen samples collected.
Protein Content - Change in Plasma Protein Levels | Intervention Trial at the 190 minute mark
  Assessment of plasma protein levels within biospecimen samples collected.
Protein Content - Change in Plasma Protein Levels | Intervention Trial at the 220 minute mark
  Assessment of plasma protein levels within biospecimen samples collected.
Protein Content - Change in Plasma Protein Levels | Rehydration Protocol - 24 hours post-intervention
  Assessment of plasma protein levels within biospecimen samples collected.
Hydration Status - Change in Acute Urine Color | Phase-specific PRE Session
  Assessment of kidney function via urine biomarkers collected during data procedures.
Hydration Status - Change in 24-h Urine Color | Phase-specific PRE Session
  Assessment of kidney function via urine biomarkers collected during data procedures.
Hydration Status - Change in Acute Urine Color | Intervention Trial at the -45 minute mark
  Assessment of kidney function via urine biomarkers collected during data procedures.
Hydration Status - Change in 24-h Urine Color | Intervention Trial at the -45 minute mark
  Assessment of kidney function via urine biomarkers collected during data procedures.
Hydration Status - Change in Urine Color | Intervention Trial at the 0 minute mark
  Assessment of kidney function via urine biomarkers collected during data procedures.
Hydration Status - Change in Urine Color | Intervention Trial at the 40 minute mark
  Assessment of kidney function via urine biomarkers collected during data procedures.
Hydration Status - Change in Urine Color | Intervention Trial at the 80 minute mark
  Assessment of kidney function via urine biomarkers collected during data procedures.
Hydration Status - Change in Urine Color | Intervention Trial at the 220 minute mark
  Assessment of kidney function via urine biomarkers collected during data procedures.
Hydration Status - Change in Urine Color | Rehydration Protocol - 3 hours post-intervention
  Assessment of kidney function via urine biomarkers collected during data procedures.
Hydration Status - Change in Urine Color | Rehydration Protocol - 6 hours post-intervention
  Assessment of kidney function via urine biomarkers collected during data procedures.
Hydration Status - Change in Urine Color | Rehydration Protocol - 15 hours post-intervention
  Assessment of kidney function via urine biomarkers collected during data procedures.
Hydration Status - Change in Urine Color | Rehydration Protocol - 24 hours post-intervention
  Assessment of kidney function via urine biomarkers collected during data procedures.
Cardiovascular Function - Change in Blood Pressure | Phase-specific PRE Session
  Assessment of cardiovascular function via blood pressure changes during data collection procedures
Cardiovascular Function - Change in Blood Pressure | Intervention Trial at the -45 minute mark
  Assessment of cardiovascular function via blood pressure changes during data collection procedures
Cardiovascular Function - Change in Blood Pressure | Intervention Trial at the 0 minute mark
  Assessment of cardiovascular function via blood pressure changes during data collection procedures
Cardiovascular Function - Change in Blood Pressure | Intervention Trial at the 40 minute mark
  Assessment of cardiovascular function via blood pressure changes during data collection procedures
Cardiovascular Function - Change in Blood Pressure | Intervention Trial at the 80 minute mark
  Assessment of cardiovascular function via blood pressure changes during data collection procedures
Cardiovascular Function - Change in Blood Pressure | Intervention Trial at the 220 minute mark
  Assessment of cardiovascular function via blood pressure changes during data collection procedures
Cardiovascular Function - Change in Blood Pressure | Rehydration Protocol - 24 hours post-intervention
  Assessment of cardiovascular function via blood pressure changes during data collection procedures
Cardiovascular Function - Change in Heart Rate Variability | Phase-specific PRE Session
  Assessment of cardiovascular function via HRV changes during data collection procedures
Cardiovascular Function - Change in Heart Rate Variability | Intervention Trial at the -45 minute mark
  Assessment of cardiovascular function via HRV changes during data collection procedures
Cardiovascular Function - Change in Heart Rate Variability | Intervention Trial at the 0 minute mark
  Assessment of cardiovascular function via HRV changes during data collection procedures
Cardiovascular Function - Change in Heart Rate Variability | Intervention Trial at the 40 minute mark
  Assessment of cardiovascular function via HRV changes during data collection procedures
Cardiovascular Function - Change in Heart Rate Variability | Intervention Trial at the 80 minute mark
  Assessment of cardiovascular function via HRV changes during data collection procedures
Cardiovascular Function - Change in Heart Rate Variability | Intervention Trial at the 220 minute mark
  Assessment of cardiovascular function via HRV changes during data collection procedures
Cardiovascular Function - Change in Heart Rate Variability | Rehydration Protocol - 24 hours post-intervention
  Assessment of cardiovascular function via HRV changes during data collection procedures
Cognitive Differences - Changes in 2 Choice Reaction Time | Intervention Trial at -45 minute mark
  This test will be used for the assessment of attention and processing speed when presented with the opportunity to make a simple choice. The test will include a "*" or "o" which will be presented on the computer screen display. The participant will be instructed to respond as quickly as possible by pressing the designated button for each stimulus as it appears on the screen.
Cognitive Differences - Changes in 2 Choice Reaction Time | Intervention Trial at 80 minute mark
  This test will be used for the assessment of attention and processing speed when presented with the opportunity to make a simple choice. The test will include a "*" or "o" which will be presented on the computer screen display. The participant will be instructed to respond as quickly as possible by pressing the designated button for each stimulus as it appears on the screen.
Cognitive Differences - Changes in 2 Choice Reaction Time | Intervention Trial at 220 minute mark
  This test will be used for the assessment of attention and processing speed when presented with the opportunity to make a simple choice. The test will include a "*" or "o" which will be presented on the computer screen display. The participant will be instructed to respond as quickly as possible by pressing the designated button for each stimulus as it appears on the screen.
Cognitive Differences - Changes in 2 Choice Reaction Time | Rehydration Protocol - 24 hours post-intervention
  This test will be used for the assessment of attention and processing speed when presented with the opportunity to make a simple choice. The test will include a "*" or "o" which will be presented on the computer screen display. The participant will be instructed to respond as quickly as possible by pressing the designated button for each stimulus as it appears on the screen.
Cognitive Differences - Changes in Stroop Test | Intervention Trial at the -45 minute mark
  This test will be used for the assessment of processing speed, selective attention, interference, and executive functioning skills by correctly identifying either the word- or color-based stimuli presented on the computer screen.
Cognitive Differences - Changes in Stroop Test | Intervention Trial at the 80 minute mark
  This test will be used for the assessment of processing speed, selective attention, interference, and executive functioning skills by correctly identifying either the word- or color-based stimuli presented on the computer screen.
Cognitive Differences - Changes in Stroop Test | Intervention Trial at the 220 minute mark
  This test will be used for the assessment of processing speed, selective attention, interference, and executive functioning skills by correctly identifying either the word- or color-based stimuli presented on the computer screen.
Cognitive Differences - Changes in Stroop Test | Rehydration Protocol - 24 hours post-intervention
  This test will be used for the assessment of processing speed, selective attention, interference, and executive functioning skills by correctly identifying either the word- or color-based stimuli presented on the computer screen.
Cognitive Differences - Changes in Matching to Samples Test | Intervention Trial at the -45 minute mark
  This test will be used for the assessment of spatial processing and visuo-spatial working memory by correctly identifying the correct sample pattern when presented with a comparison of a similar grid on the computer screen.
Cognitive Differences - Changes in Matching to Samples Test | Intervention Trial at the 80 minute mark
  This test will be used for the assessment of spatial processing and visuo-spatial working memory by correctly identifying the correct sample pattern when presented with a comparison of a similar grid on the computer screen.
Cognitive Differences - Changes in Matching to Samples Test | Intervention Trial at the 220 minute mark
  This test will be used for the assessment of spatial processing and visuo-spatial working memory by correctly identifying the correct sample pattern when presented with a comparison of a similar grid on the computer screen.
Cognitive Differences - Changes in Matching to Samples Test | Rehydration Protocol - 24 hours post-intervention
  This test will be used for the assessment of spatial processing and visuo-spatial working memory by correctly identifying the correct sample pattern when presented with a comparison of a similar grid on the computer screen.
Performance Differences - Changes in Balance | Intervention Trial at -45 minute mark
  Participants will be evaluated for balance capabilities through use of the BESS test.
Performance Differences - Changes in Balance | Intervention Trial at 80 minute mark
  Participants will be evaluated for balance capabilities through use of the BESS test.
Performance Differences - Changes in Balance | Intervention Trial at 220 minute mark
  Participants will be evaluated for balance capabilities through use of the BESS test.
Performance Differences - Changes in Balance | Rehydration Protocol - 24 hours post-intervention
  Participants will be evaluated for balance capabilities through use of the BESS test.
Performance Differences - Changes in Muscular Strength Testing | Intervention Trial at the -45 minute mark
  Participants will be evaluated for grip strength via implementation of a hand-held dynamometer.
Performance Differences - Changes in Muscular Strength Testing | Intervention Trial at the 80 minute mark
  Participants will be evaluated for grip strength via implementation of a hand-held dynamometer.
Performance Differences - Changes in Muscular Strength Testing | Intervention Trial at the 220 minute mark
  Participants will be evaluated for grip strength via implementation of a hand-held dynamometer.
Performance Differences - Changes in Muscular Strength Testing | Rehydration Protocol - 24 hours post-intervention
  Participants will be evaluated for grip strength via implementation of a hand-held dynamometer.
Performance Differences - Changes in Muscular Endurance Testing | Intervention Trial at the -45 minute mark
  Participants will be evaluated for grip strength endurance via implementation of a hand-held dynamometer.
Performance Differences - Changes in Muscular Endurance Testing | Intervention Trial at the 80 minute mark
  Participants will be evaluated for grip strength endurance via implementation of a hand-held dynamometer.
Performance Differences - Changes in Muscular Endurance Testing | Intervention Trial at the 220 minute mark
  Participants will be evaluated for grip strength endurance via implementation of a hand-held dynamometer.
Performance Differences - Changes in Oxygen Consumption | Intervention Trial at the 100 minute mark
  Participants will be evaluated for oxygen consumption while performing exercise at approximately 40% of velocity obtained during their previously measured VO2max test. These assessments will be completed in 5 minute intervals during the Intervention Trials.
Performance Differences - Changes in Oxygen Consumption | Intervention Trial at the 160 minute mark
  Participants will be evaluated for oxygen consumption while performing exercise at approximately 40% of velocity obtained during their previously measured VO2max test. These assessments will be completed in 5 minute intervals during the Intervention Trials.
Performance Differences - Changes in Oxygen Consumption | Intervention Trial at the 215 minute mark
  Participants will be evaluated for oxygen consumption while performing exercise at approximately 40% of velocity obtained during their previously measured VO2max test. These assessments will be completed in 5 minute intervals during the Intervention Trials.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas J Casa, PhD, Principal Investigator — Korey Stringer Institute - UConn
Locations (1):
- Korey Stringer Institute at the University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No